CLINICAL TRIAL: NCT06995430
Title: A Phase 3b, Open-Label, Multi-Center Study to Assess the Immune Response And Safety of The Meningococcal Group B Vaccine Rmenb+Omv Nz When Administered to Healthy Participants Aged 10 To 20 Years Old, Who Were Primed During the First 2 Years Of Life
Brief Title: A Phase 3 Study to Assess the Immune Response And Safety Of Rmenb+Omv Nz In Primed Healthy Participants (10 To 20 Years Old)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 220030; 2024-519549-31 (EudraCT Number)
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Meningitis
Keywords: Meningitis; booster dose; Bexsero; Immune response
MeSH Terms: conditions — Meningitis | interventions — 4CMenB vaccine

STUDY DESIGN:
Masking Description: This is an Open-Label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primed group (Experimental): Participants who were primed with rMenB+OMV NZ in a 2+1 or 3+1 schedule during the first 2 years of life will receive 1 dose of rMenB+OMV NZ at Day 1.
  Interventions: Biological: rMenB+OMV NZ vaccine
- Naive group (Active Comparator): Participants who are group B-meningococcal-vaccine-naive within the same age range as the primed group receive 2 doses of rMenB+OMV NZ at Day 1 and Day 31.
  Interventions: Biological: rMenB+OMV NZ vaccine

INTERVENTIONS:
Biological: rMenB+OMV NZ vaccine — 1 dose in the Primed group or 2 doses in the Naive group.
  Other Names: Bexsero

SUMMARY:
The main purpose of this study is to evaluate the immune response and safety of a booster dose of the meningococcal group B vaccine, rMenB+OMV NZ (also known as Bexsero), in adolescents and young adults aged 10 to 20 years. This study focuses on individuals who were first vaccinated with rMenB+OMV NZ as infants. The primary hypothesis is that a booster dose of the vaccine will elicit a stronger immune response in these primed individuals compared to those who have never received any group B meningococcal vaccine, referred to as 'nave' participants.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

For primed group only:

• Participated who were primed with rMenB + OMV NZ in only either 3+1 or 2+1 schedule during the first 2 years of life as confirmed by electronic or paper vaccination record.

OR

For naïve group only:

• Electronic or paper vaccination record confirmed participant who has never received any group B meningococcal vaccine and is recruited in the same country as primed participants.

For all participants:

* Participants and/or participants' parent(s)/ legally acceptable representative(s) (LAR[s]), who, in the opinion of the investigator, can and will comply with the requirements of the protocol
* Written or witnessed/thumb printed informed consent obtained from the participant / parent(s)/LAR(s) of the participant prior to performance of any study-specific procedure.
* Written informed assent obtained from the participant (if applicable) along with informed consent from the participant's parent(s)/LAR(s) prior to performing any study specific procedure.

Note: For age 10-16 years, parents or LAR to give consent along with participants, based on country regulations for participants and for >16/18 to 20 years, participants give consent independent of parents/LARs, or as per local country regulations.

* A male or female between, and including, 10 and 20 years of age at the time of the first study intervention administration.
* Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, hysterectomy, bilateral ovariectomy.
* Female participants of childbearing potential may be enrolled in the study, if the participant:

  * has practiced adequate contraception for 1 month prior to study intervention administration, and
  * has a negative pregnancy test on the day of study intervention administration, and
  * has agreed to continue adequate contraception during the entire study treatment period.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Medical conditions

* Current or previous, confirmed or suspected disease caused by N. meningitidis.
* Known exposure to an individual with laboratory confirmed N. meningitidis infection, within 60 days prior to enrollment.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention.
* Medical conditions representing a contraindication to intramuscular vaccination and blood draws.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.

Prior/Concomitant therapy

* Use of any investigational or non-registered product (drug, vaccine or medical device) other than the study intervention during the period beginning 30 days before the first dose of study intervention (Day -29 to Day 1), or their planned use during the study period.
* Chronic administration of immune-modifying drugs (defined as more than 14 consecutive days in total) and/or planned use of long-acting immune-modifying treatments at any time up to the end of the study.

  * Within 90 days prior to study intervention administration: for corticosteroids, this will mean prednisone equivalent ≥20 mg/day for adult participants or >= 0.5 mg/kg/day with maximum of 20 milligram (mg)/day for pediatric participants. Inhaled and topical steroids are allowed.
  * Within 90 days prior to study intervention administration: long-acting immune-modifying drugs including among others immunotherapy (e.g., TNF-inhibitors), monoclonal antibodies, antitumoral medication.
* Administration of immunoglobulins and/or any blood products or plasma derivatives within 180 days prior to study intervention administration and/or planned use at any time up to the end of the study.

For primed group only:

• Participants who received additional dose(s) of group B meningococcal vaccine other than 2+1 or 3+1 schedule prior to study intervention administration.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug/vaccine/invasive medical device).

Other exclusion criteria

* Pregnant or lactating female participant.
* Any study personnel or their immediate dependents, family, or household member.
* Child in care.

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 226 (Actual)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
hSBA Geometric mean titers (GMTs) ratio against each MenB indicator strain | At Day 31

SECONDARY OUTCOMES:
Number of participants with hSBA titers greater than or equal (>=) to pre-defined limit of detection against each MenB indicator strain | At Day 31
Number of participants with hSBA titers >= lower limit of quantification (LLOQ) against each MenB indicator strain | At Day 31
Number of participants with four-fold increase in hSBA titers | At Day 31
hSBA GMTs against each MenB indicator strain | At Day 31 compared to Day 1
hSBA Geometric Mean Ratios (GMRs) against each MenB indicator strain | At Day 31 compared to Day 1
Number of participants with hSBA titers >= to pre-defined limit of detection against each MenB indicator strain | At Day 1
Number of participants with hSBA titers >= LLOQ against each MenB indicator strain | At Day 1
hSBA GMTs against each MenB indicator strain | At Day 1
Number of participants with solicited administration site events | Day 1 (day of injection) to Day 7
  The solicited administration site events include injection site pain, erythema (redness), swelling and induration.
Number of participants with solicited systemic events | Day 1 (day of injection) to Day 7
  The solicited systemic events include fever (temperature >= 38.0°C), headache, myalgia (muscle pain), arthralgia (joint pain), fatigue (tiredness), nausea.
Number of participants with any unsolicited adverse events (AEs) | Day 1 (day of injection) to Day 31
Number of participants with adverse events of special interest (AESI): arthritis, serious adverse events (SAEs), AEs leading to withdrawal | Day 1 to Day 31 (throughout the study period)

CONTACTS AND LOCATIONS:
Locations (17):
- Finland (8):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- Italy (4):
  - GSK Investigational Site, Florence
  - GSK Investigational Site, Genova
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Novara
- Spain (2):
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
- United Kingdom (3):
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, London
  - GSK Investigational Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf